CLINICAL TRIAL: NCT05148494
Title: Transanal Endoscopic Surgery: a Randomized Controlled Trial Comparing Fleet Enema vs Oral Mechanical Bowel Prep (TESEO Trial)
Brief Title: TES RCT Fleet Enema vs Oral Mechanical Bowel Prep
Acronym: TESEO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Katerina Neumann, Assistant Professor, colorectal surgeon, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Protocol v2
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Neoplasms; Surgery
Keywords: transanal endoscopic surgery; TEM; TAMIS; rectal neoplasm; oral mechanical bowel preparation; fleet enema; Ottawa bowel prep score
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — sodium phosphate; Pico-Salax

STUDY DESIGN:
Intervention Model Description: A single center, 2-arm, single blinded randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant will receive information pertaining to which arm of the trial they have been randomized to by the research coordinator. The surgeons, residents, any other physicians involved in the care of the patient, and nursing staff will all be blinded to the treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fleet Enema (Active Comparator): Patient is to administer one sodium bisphosphate (Fleet) enema at home 2 hours prior to arrival for surgery and a second enema one hour prior to arrival for surgery. Each 120 mL application of rectally administered enema contains 19g of monobasic sodium phosphate and 9 g of dibasic sodium phosphate. Patient is to follow standard packaging instructions from the manufacturer.
  Interventions: Drug: Fleet Enema
- Pico Salax (Active Comparator): Patient is to take Pico Salax oral bowel preparation which is a combination product consisting of 10 mg picosulfate sodium, 3.5 g magnesium oxide, and 12 g citric acid per sachet the day prior to surgery. Patient is to take 2 doses of this product, as per standard packaging instructions from the manufacturer. Specifically patient is to take the first packet contents dissolved in 150 mL water at 3pm the day before surgery. Patient is to take the second packet dissolved in 150 mL water at 8pm the day before surgery. Patient should drink 2-3L of clear liquids after each dose, for a total of 4-6L.
  Interventions: Drug: Pico-Salax

INTERVENTIONS:
Drug: Fleet Enema — standard pre-op application, see arm description
  Arms: Fleet Enema
Drug: Pico-Salax — standard pre-op application, see arm description
  Arms: Pico Salax

SUMMARY:
There is no consensus about the best bowel preparation prior to transanal endoscopic surgery TES). Cleanliness and visibility in the rectosigmoid and rectum are of utmost importance, possibly even more so than during colonoscopy, to facilitate safe, precise and efficient resection of the rectal lesion and potentially adequate closure of the defect. Both Fleet enemas and oral mechanical bowel preparation are considered standard of care in preparation for TES. This single center two arm single blinded randomized controlled trial will compare the effectiveness of Fleet enemas in comparison to Pico Salax oral mechanical bowel preparation in cleansing the rectum as measured by a modified version of the Ottawa Bowel Prep Scale.

DETAILED DESCRIPTION:
Oral mechanical bowel preparation with Pico Salax (picosulfate sodium, magnesium oxide, and citric acid) or alternative is considered a standard modality for cleansing the entire colon prior to colonoscopy or surgical procedures. Fleet enemas are sodium phosphate-based laxatives in the form of a liquid inserted rectally, which are also very effective at evacuating the solid stool from the sigmoid and rectum in preparation for procedures such as flexible sigmoidoscopy or anoscopy, which only require visualization of the distal colon and rectum. Commonly, endoscopists use the well validated bowel preparation scores such as the Boston Bowel Prep Score, Aronchick Scale or the Ottawa Bowel Prep Scale when evaluating the effectiveness of such bowel preparation regimens at clearing away all debris and opaque liquid from the colon. Few studies have been performed to evaluate whether an oral mechanical bowel preparation or a rectal application by means of fleet enemas or alternatives gives better visibility or is preferred by the patient. A randomized controlled trial comparing two fleet enemas with an oral preparation that consisted of magnesium citrate and two Dulcolax tablets for flexible sigmoidoscopy, were able to show that patient acceptance, encounter time, technical ease, quality of colon preparation was significantly better with the oral form of colon preparation than with standard fleet enemas. On the other hand, another randomized controlled trial were able to show that fleet enemas were superior to picosulfate based oral bowel preparation for flexible sigmoidoscopy while also showing a decreased incidence of associated adverse symptoms, and better patient tolerance. Conflicting studies exist. Both bowel regimens are considered standard of care in preparation for surgery of the sigmoid and rectum. Fleet enemas seem to be the preparation most commonly used for flexible sigmoidoscopy.

Transanal endoscopic surgery (TES) is a minimally invasive technique used to perform full thickness excisions of rectal lesions (benign and malignant) with precision, allowing access to lesions in the rectum as high as 22 cm from the anus. The technique can be performed using either the rigid transanal endoscopic microsurgery (TEM) platform or the flexible port termed transanal endoscopic minimally invasive surgery (TAMIS). The technique decreases risk of positive margins and local recurrence in comparison to standard local excision techniques in the operating room. It is the preferred method of local excision of rectal lesions. As with polyp detection and removal during flexible sigmoidoscopy, TES for rectal neoplasms requires excellent visibility and minimization of debris in order to be able to perform the precise excision of the lesion and help facilitate closure of the full thickness defect in the rectal wall. TES is performed globally with no consensus about the optimal bowel preparation regimen for achieving visibility and facilitating the easiest, most efficient and safest dissection.

Objectives:

The primary objective of this study is to determine whether oral Pico Salax bowel preparation regimen achieves a higher score on the Ottawa Bowel Prep Scale specifically for the rectosigmoid segment in comparison to 2 fleet enemas during TES.

The secondary objectives include validation of the Ottawa Bowel Prep Scale specifically for use with fleet enemas or Pico Salax for the rectosigmoid segment during TES; determining if there are differences in length of time spent cleaning the operative field by the surgeon; the ability to close the defect; post-operative short-term complications, and patient tolerability of the preparation.

This study will serve as a pilot study for a potentially larger multi-center pan Canadian RCT. The TEMPEST group is a collaboration of TES trained surgeons across Canada at tertiary care teaching hospitals, involved in research collaborations. The results of this study will be used to see if randomization to two different bowel regimens in this very select group of patients undergoing trans-anal surgery is feasible and can yield informative data. The study will be powered for the primary objective, but we will be collecting data on numerous secondary objectives which may show important trends. If the study proves to be feasible, the next step would be to expand the study to several other centers across Canada as part of the TEMPEST collaborative, in order to collect much larger datasets and the power to look much more closely at not only the primary objective but also the secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* undergoing transanal endoscopic surgery at the QEII Health Sciences Center in Halifax by one of the colorectal trained surgeons

Exclusion Criteria:

* chronic constipation not well controlled with diet or stool softening agents
* previous pelvic radiation
* inflammatory bowel disease
* repeat transanal surgery for the same lesion
* patient unable to self-administer enemas
* patient unable to tolerate either of the 2 bowel preps due to medical reasons
* age over 75
* clear diagnosis of congestive heart failure
* daily use of Lasix or similar loop diuretic
* chronic steroid use
* Transanal Endoscopic Surgery combined with another surgical procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Quality of bowel preparation | A one-time intra-operative assessment for each patient
  Measurement of the quality of cleanse of the rectum, expressed as a score on a modified version of the Ottawa Bowel Prep Scale (OBPS).
  The OBPS will be used to assess the one segment of the bowel visualized during TES surgery (rectosigmoid) using the segmental scale 0-4, where 0 is the best score and 4 is inadequate.

SECONDARY OUTCOMES:
Validation of the modified version of the Ottawa Bowel Prep Scale | A one-time intra-operative assessment for each patient by a second blinded surgeon
  validation of the modified version of the OBPS as it applies to the use of Fleet enema and Pico Salax oral bowel prep in the rectosigmoid segment specifically for use in preparation for TES
Time spent cleaning operating field | A one-time intra-operative assessment for each patient
  A measure of the time spent cleansing the operating field by the surgeon as per review of recording of the surgery
Ability to close the surgical defect | A one-time intra-operative assessment for each patient
  An assessment as to whether the surgical wound in the rectum was left open or sutured closed
Patient tolerability of preparation | A one-time pre-op assessment for each patient the morning of surgery
  An assessment of the patients tolerability of the prep, symptoms associated with the prep, whether they were able to complete the prep, satisfaction and willingness to take the same prep in the future, performed using a questionnaire. In the questionnaire, the severity of the symptoms associated with the prep can be selected from mild, moderate, severe, and intolerable.
Post-operative complications | At discharge and at 6 weeks post-operatively
  An assessment of in-hospital as well as short term complications assessed at time of discharge and during 6-week post-operative visit

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Neumann, Principal Investigator — NSHA
Locations (1):
- Victoria General Hospital, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Parekh PJ, Oldfield EC 4th, Johnson DA. Bowel preparation for colonoscopy: what is best and necessary for quality? Curr Opin Gastroenterol. 2019 Jan;35(1):51-57. doi: 10.1097/MOG.0000000000000494. PMID 30489414
- [Background] Parra-Blanco A, Ruiz A, Alvarez-Lobos M, Amoros A, Gana JC, Ibanez P, Ono A, Fujii T. Achieving the best bowel preparation for colonoscopy. World J Gastroenterol. 2014 Dec 21;20(47):17709-26. doi: 10.3748/wjg.v20.i47.17709. PMID 25548470
- [Background] Atkin WS, Hart A, Edwards R, Cook CF, Wardle J, McIntyre P, Aubrey R, Baron C, Sutton S, Cuzick J, Senapati A, Northover JM. Single blind, randomised trial of efficacy and acceptability of oral picolax versus self administered phosphate enema in bowel preparation for flexible sigmoidoscopy screening. BMJ. 2000 Jun 3;320(7248):1504-8; discussion 1509. doi: 10.1136/bmj.320.7248.1504. PMID 10834891
- [Background] Ruangsin S, Chowchuvech V. A randomized double-blind controlled trial comparing two forms of enema for flexible sigmoidoscopy. J Med Assoc Thai. 2007 Nov;90(11):2296-300. PMID 18181310
- [Background] Preston KL, Peluso FE, Goldner F. Optimal bowel preparation for flexible sigmoidoscopy--are two enemas better than one? Gastrointest Endosc. 1994 Jul-Aug;40(4):474-6. doi: 10.1016/s0016-5107(94)70213-6. PMID 7926539
- [Background] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102
- [Background] Calderwood AH, Jacobson BC. Comprehensive validation of the Boston Bowel Preparation Scale. Gastrointest Endosc. 2010 Oct;72(4):686-92. doi: 10.1016/j.gie.2010.06.068. PMID 20883845
- [Background] Aronchick C, Lipschultz W, Wright S. Validation of an instrument to assess colon cleansing. Am J Gastroenterol 1993;94:2667.
- [Background] Rostom A, Jolicoeur E. Validation of a new scale for the assessment of bowel preparation quality. Gastrointest Endosc. 2004 Apr;59(4):482-6. doi: 10.1016/s0016-5107(03)02875-x. PMID 15044882
- [Background] Kao D, Lalor E, Sandha G, Fedorak RN, van der Knoop B, Doornweerd S, van Kooten H, Schreuders E, Midodzi W, Veldhuyzen van Zanten S. A randomized controlled trial of four precolonoscopy bowel cleansing regimens. Can J Gastroenterol. 2011 Dec;25(12):657-62. doi: 10.1155/2011/486084. PMID 22175055
- [Background] Holt EW, Yimam KK, Ma H, Shaw RE, Sundberg RA, Verhille MS. Patient tolerability of bowel preparation is associated with polyp detection rate during colonoscopy. J Gastrointestin Liver Dis. 2014 Jun;23(2):135-40. doi: 10.15403/jgld.2014.1121.232.ewh1. PMID 24949604
- [Background] Kim MJ, Hong CW, Kim BC, Park SC, Han KS, Joo J, Oh JH, Sohn DK. Phase II Randomized Controlled Trial of Combined Oral laxatives Medication for BOwel PREParation (COMBO-PREP study). Medicine (Baltimore). 2016 Feb;95(7):e2824. doi: 10.1097/MD.0000000000002824. PMID 26886637
- [Background] Sharma VK, Chockalingham S, Clark V, Kapur A, Steinberg EN, Heinzelmann EJ, Vasudeva R, Howden CW. Randomized, controlled comparison of two forms of preparation for screening flexible sigmoidoscopy. Am J Gastroenterol. 1997 May;92(5):809-11. PMID 9149190
- [Background] Drew PJ, Hughes M, Hodson R, Farouk R, Lee PW, Wedgwood KR, Monson JR, Duthie GS. The optimum bowel preparation for flexible sigmoidoscopy. Eur J Surg Oncol. 1997 Aug;23(4):315-6. doi: 10.1016/s0748-7983(97)90723-x. PMID 9315059
- [Background] Bini EJ, Unger JS, Rieber JM, Rosenberg J, Trujillo K, Weinshel EH. Prospective, randomized, single-blind comparison of two preparations for screening flexible sigmoidoscopy. Gastrointest Endosc. 2000 Aug;52(2):218-22. doi: 10.1067/mge.2000.107907. PMID 10922094
- [Background] Fincher RK, Osgard EM, Jackson JL, Strong JS, Wong RK. A comparison of bowel preparations for flexible sigmoidoscopy: oral magnesium citrate combined with oral bisacodyl, one hypertonic phosphate enema, or two hypertonic phosphate enemas. Am J Gastroenterol. 1999 Aug;94(8):2122-7. doi: 10.1111/j.1572-0241.1999.01308.x. PMID 10445538